CLINICAL TRIAL: NCT00902642
Title: Does Training in Psychosocial Methods for Treatment Providers Improve Outcome for Pain Patients at Risk of Long-Term Disability? A Randomised Controlled Trail of a Course for Physical Therapists
Brief Title: What is the Effect of a Course for Treatment Providers on Their Patient Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Örebro University, Sweden (Other); School of Law, Psychology, and Social Work, Örebro University, Sweden (Unknown)
Responsible Party: Steven J Linton, Ph. D., Professor of Clinical Psychology, Center for Health and Medical Psychology and School of Law, Psychology, and Social Work, Örebro University, Sweden
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M-127
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Pain
Keywords: Physical therapy,; musculoskeletal pain,; psychosocial factors,; dissimilation,; evidence based,; education
MeSH Terms: conditions — Pain; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention)
- Course on psychosocial factors (Active Comparator): an eight day university training course for physical therapists designed to integrating psychosocial factors in clinical practice on a patient level
  Interventions: Behavioral: an eight day university training course designed to integrating psychosocial factors in clinical practice on a patient level

INTERVENTIONS:
Behavioral: an eight day university training course designed to integrating psychosocial factors in clinical practice on a patient level — an eight day university training course on psychosocial factors for physical therapists
  Arms: Course on psychosocial factors

SUMMARY:
The goal is to acquire more in-depth knowledge on physical therapists' attitudes towards and beliefs about psychosocial factors in back pain, how physical therapists integrate psychosocial factors into their clinical practice and the effects of a training program for physical therapists in psychosocial factors on clinical practice and thereby on patient outcome in terms of disability, pain, catastrophizing, and treatment satisfaction.

DETAILED DESCRIPTION:
Neck and back pain continue to be extremely common, with a high prevalence and wide socio-economic consequences all over the industrialized world. Through the years a growing interest has risen for other factors than the pure biomedical or biomechanical. This has led to a new clinical model for the treatment of back pain; the biopsychosocial model of illness. Treatment based on the biopsychosocial model not only must address the biological basis of symptoms, but must incorporate the full range of social and psychological factors that have been shown to affect pain, distress and disability.

Since there is today strong evidence indicating that psychosocial factors have a greater impact on disability then biomechanical or biomedical factors and strong evidence that psychosocial factors are strongly linked to the transition from acute to chronic pain, concept of psychosocial risk factors has been developed. Although the concept of psychosocial risk factors still is relatively new, there seems to be an international consensus about the importance of psychosocial risk factors for the prevention of the development of chronic pain but there appears to be considerable uncertainty about the clinical application.

Health care providers' (HCPs') attitudes and beliefs appear to influence the information they provide to patients. This may subsequently result in different patient outcome depending on the HCPs' attitudes and beliefs. Physical therapists attitudes and beliefs are relatively unexplored but seem to have an effect on patients' attitudes and beliefs, which can affect patient outcome in terms of sick leave, health care use and function.

HCP attitudes and beliefs towards psychosocial factors are relatively unexplored. Yet, it seems physical therapists do not necessarily accept new evidence-based information and may have difficulties in applying evidence-based information in their clinical practice. Implementation and dissemination of evidence-based psychosocial factors requires favourable attitudes, knowledge and skills to ensure a behavioural change on behave of the physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Musculoskeletal pain,
* Age between 18 and 65

Exclusion Criteria:

* Sick leave for more than 3 months during the past year as a result of present the musculoskeletal pain problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Disability | treatment start and 6 month follow up

SECONDARY OUTCOMES:
catastrophizing | treatment start and 6 month follow up
treatment satisfaction | 6 month follow up
satisfaction with treatment result | 6 month follow up
Pain | treatment start and 6 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Linton, PH.D., Study Director — Center for Health and Medical Psychology and School of Law, Psychology, and Social Work, Örebro University, Sweden
Locations (1):
- Mälardalens högskola, Eskilstuna, Sweden

REFERENCES:
- [Derived] Overmeer T, Boersma K, Denison E, Linton SJ. Does teaching physical therapists to deliver a biopsychosocial treatment program result in better patient outcomes? A randomized controlled trial. Phys Ther. 2011 May;91(5):804-19. doi: 10.2522/ptj.20100079. Epub 2011 Mar 30. PMID 21451098